CLINICAL TRIAL: NCT06084455
Title: The Effect of Aerobic Exercise on Brain Connectivity
Brief Title: TMS-evoked Potentials During Aerobic Exercise
Acronym: TMS-EEGxercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Enrico De Martino, Dr, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20210047-4
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2023-10

CONDITIONS: Transcranial Magnetic Stimulation; Electroencephalography; Aerobic Exercise
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aerobic exercise (Experimental): 30 minutes of aerobic exercise will be performed by the participants before and after cortical connectivity measurements.
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Aerobic exercise — 30 minutes of aerobic exercise on a stationary bike

SUMMARY:
This study investigates the modification of the local-to-global connectivity pattern in response to a session of aerobic exercise. Transcranial magnetic stimulation (TMS) will be applied to elicit electroencephalography (EEG) responses in healthy volunteers. The TMS-evoked potentials (TEPs) will be recorded and serve as a reflection of cortical reactivity and connectivity to TMS.

DETAILED DESCRIPTION:
Chronic musculoskeletal pain disorders rank second only to mental and behavioural disorders as a major contributor to worldwide years lived with disability. Chronic musculoskeletal pain restricts mobility, decreases cardiorespiratory capacity and musculoskeletal function, and ultimately reduces exercise capacity and quality of life. Thus, there is an urgent need for new, effective, and affordable strategies to address this growing problem, particularly in health systems around the world.

Abnormal brain connectivity patterns disrupt normal brain function in a specific neural network, causing brain circuit malfunctions and resulting in symptoms such as chronic pain. The advent of electroencephalography (EEG) compatible with transcranial magnetic stimulation (TMS-EEG) has allowed the measurement of the cortical excitability and connectivity of a single pulse of TMS in any scalp region, providing insights into cortical excitability and connectivity that were not previously possible with techniques exclusively based on MEP, create a map of activation caused by a localized pulse of stimulation. Furthermore, TMS-EEG allows recording the spread and the characteristics of the perturbations caused by a single TMS pulse across the cortex (recorded by several electrodes from an EEG cap). Physical exercise has been shown to have a positive impact on brain functioning. Regular exercise promotes the growth of new brain cells and improves the survival of existing ones. Studies have shown that regular exercise improves cognitive function, memory, and mood, and exercise has been linked to increased production of neurotransmitters, hormones, and growth factors that promote brain health. However, to date, no studies have investigated the effect of aerobic exercise on brain excitability and connectivity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Speak and understand English

Exclusion Criteria:

* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, musculoskeletal or mental illnesses
* Lack of ability to cooperate
* History of chronic pain or current acute pain
* Contraindications to rTMS application (history of epilepsy, metal in the head or jaw etc.).
* Failure to pass the "TASS questionnaire" (TASS = Transcranial Magnetic Stimulation Adult Safety Screen)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Cortical connectivity | Cortical connectivity changes will be investigated before and after 30-min aerobic exercise (1 hour)
  Global and local mean field amplitude

SECONDARY OUTCOMES:
Cortical excitability | Cortical excitability changes will be investigated before and after 30-min aerobic exercise (1 hour)
  TMS-evoked potentials

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Gistrup, North Denmark, Denmark